CLINICAL TRIAL: NCT07161349
Title: Plantar Pressure Distribution In Relation to The Way of Carrying Backpack In Adolescents
Brief Title: The Relation Between Plantar Pressure Distribution on the Foot and The Way of Carrying Backpack in Students Between 12 to 18 Years
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Amira Ibrahem, B.Sc. in Physical Therapy, Cairo University
Other Study IDs: 012/005593
Record Dates: First submitted 2025-08-30; First posted 2025-09-08 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Healthy Participants
Keywords: Plantar pressure distribution; Carrying backpack; Adolescents

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
What is this study about? This is an observational study that investigates how different ways of carrying a school backpack affect the pressure distribution on the soles of the feet (plantar pressure) in adolescents.

The main questions it aims to answer are:

Does carrying a backpack on one shoulder (unilaterally) change the pressure on the bottom of the foot compared to carrying it on both shoulders (bilaterally)?

Does carrying a backpack change the amount of the foot that touches the ground (contact area)?

Are there differences in foot pressure between the right and left foot based on how the backpack is carried?

Researchers compared four different carrying conditions to see their effects:

Carrying no backpack.

Carrying a backpack on both shoulders.

Carrying a backpack on the right shoulder only.

Carrying a backpack on the left shoulder only.

Who participated? The study included 92 healthy adolescent students (32 boys and 60 girls) from Mansoura City, Egypt. Their ages ranged from 12 to 18 years old, they had a normal Body Mass Index (BMI), and had no existing postural or musculoskeletal problems.

What did participants do?

Participants in the study were asked to:

Have their height, weight, and posture checked to ensure they are eligible.

Stand and walk barefoot on a special computerized pressure-sensitive mat (a Foot Scan Plate System).

Perform these standing and walking tasks under the four different backpack conditions listed above. The backpack was always loaded to weigh 15% of the student's body weight.

What did the study find?

The key findings were:

How you carry the backpack affects how much of your foot touches the ground. Carrying a backpack on one shoulder (especially the right) increased the contact area of both feet on the ground, both while standing and walking.

The average and maximum pressures on the soles of the feet did not change significantly. Regardless of how the backpack was carried, the intensity of the pressure under the feet remained relatively the same in these healthy adolescents.

Overall balance was maintained. Even though the carrying method changed how the feet contacted the ground, the body compensated well, and no significant imbalance in pressure between the right and left foot was found during walking.

What does this mean for patients, families, and healthcare providers?

For Teens and Families: This study highlights that how you carry your backpack matters for your foot mechanics. While a brief change may not cause immediate pain, consistently carrying a backpack on one shoulder can alter your posture and gait. It is best to use both shoulder straps to distribute weight evenly and promote healthy body alignment.

For Healthcare Providers: This research provides evidence that the backpack carriage method is a modifiable factor influencing plantar loading patterns in adolescents. Assessing a patient's backpack habits could be a useful part of evaluating complaints of foot, knee, or back pain. Educating patients and families on symmetrical load carriage and proper backpack weight (≤15% of body weight) is a valuable preventive strategy.

The bottom line: While the body can adapt to short-term uneven loading, making a habit of carrying a backpack on both shoulders is the best practice for supporting healthy foot pressure distribution and overall posture in growing adolescents.

DETAILED DESCRIPTION:
1. Abstract and Core Objective This research presents a detailed biomechanical investigation into the effects of school backpack carriage on foot function in adolescents. The study moves beyond the common focus on spinal posture to analyze the foundational segment: the foot. Utilizing advanced pedobarographic technology, it precisely measures how different loading methods-bilateral (two-strap) and unilateral (one-strap) carriage-alter the distribution of pressure across the plantar surface during static (standing) and dynamic (walking) tasks. The primary objective was to quantify these changes to inform evidence-based recommendations for preventing musculoskeletal strain in a young, developing population.
2. Background and Significance Adolescence is a period of significant skeletal and muscular development, making individuals particularly susceptible to external mechanical stresses. The ubiquitous use of backpacks, often carrying loads exceeding recommended guidelines, introduces a chronic, repetitive stressor.

   The Kinetic Chain: The human body functions as an interconnected kinetic chain. Alterations in the foundation (the feet) can have cascading effects upward, influencing ankle, knee, hip, and spinal alignment. Therefore, understanding foot pressure is crucial to understanding overall postural health.

   The Plantar Pressure Paradigm: Plantar pressure measurement is a sophisticated biomechanical tool that provides a dynamic map of force distribution. It reveals how the body adapts to load, highlighting areas of potential overloading (high pressure) or underloading, which can be precursors to pain, soft tissue damage, or long-term structural changes like flatfoot.

   The Unilateral Carriage Problem: Despite widespread knowledge of its negative effects, unilateral backpack carriage remains prevalent among adolescents due to perceived convenience and social trends. This study seeks to quantify the specific biomechanical cost of this habit.
3. Detailed Methodology 3.1. Participant Recruitment and Eligibility (Sample Demographics)

   A cohort of 92 adolescents was recruited from a mix of public and private schools in Mansoura City, Egypt, to ensure a representative sample. The stringent eligibility criteria were designed to isolate the variable of backpack carriage from other confounding factors:

   Age: 12-18 years, capturing the spectrum of pubertal growth and maturation.

   Health Status: No history of visual, vestibular, perceptual, neurological, or musculoskeletal disorders. This excluded conditions like cerebral palsy, leg length discrepancy, previous fractures, or diagnosed scoliosis beyond a minimal, normal range.

   Anthropometrics: Body Mass Index (BMI) was calculated and checked against the World Health Organization (WHO) 2007 BMI-for-age percentile charts. Only participants within the normal range (typically between the 5th and 85th percentiles) were included. This controlled for the independent influence of body weight and composition on plantar pressure.

   Postural Screening: Axial trunk rotation was measured using a scoliometer with the participant in the forward bend test position. Only those with measurements within the normal limit of 0 to 3 degrees of rotation were included, effectively screening out significant undiagnosed spinal asymmetries.

   3.2. Instrumentation and Technical Specifications

   Foot Scan Plate System (F-SCAN): This is a platform-based pressure mapping system.

   Technology: It consists of a flat, rigid plate containing a high-density grid of capacitive pressure sensors.

   Data Capture: When a subject stands or walks on the plate, each sensor measures vertical force. The system software collects this data at a high frequency (typically hundreds of Hertz), creating a dynamic, frame-by-frame image of the pressure distribution.

   Output Metrics: The system's software automatically calculates numerous parameters. This study focused on three key ones for each foot:

   Surface Contact Area (cm²): The total area of the foot in contact with the ground.

   Average Pressure (kPa): The mean force per unit area across the entire foot imprint.

   Peak (Maximum) Pressure (kPa): The highest pressure value recorded by a single sensor element, indicating a focal point of stress.

   Scoliometer: A validated, non-invasive inclinometer used to measure the angle of trunk rotation (ATR), a key indicator for scoliosis screening.

   Backpacks and Load Configuration: Two standard student backpacks were used: a double-strap model and a single-strap model. Both were simple, soft-fabric designs without internal frames or hip belts, representing a typical student backpack. The load was standardized at 15% of each participant's body weight using calibrated sandbags, a weight based on previous ergonomic studies (e.g., Chow et al., 2010) shown to induce measurable postural changes.

   3.3. Experimental Protocol and Data Collection

   The testing protocol was meticulously standardized:

   Familiarization: Participants were allowed to familiarize themselves with the laboratory setting and the pressure plate.

   Calibration: The F-SCAN system was calibrated according to manufacturer specifications before each testing session.

   Testing Conditions: Each participant was tested under four conditions in a randomized order to prevent bias:

   Condition 1 (Control): No backpack (unloaded).

   Condition 2: Backpack worn bilaterally (on both shoulders).

   Condition 3: Backpack worn unilaterally on the right shoulder.

   Condition 4: Backpack worn unilaterally on the left shoulder.

   Task Execution:

   Static Trial: Participants stood motionless on the pressure plate, looking straight ahead, with arms relaxed by their sides. Data was collected over a stable several-second interval.

   Dynamic Trial: Participants walked at a self-selected, comfortable speed across the pressure plate, capturing multiple steps. The mean value of several successful steps was used for analysis to ensure reliability.

   Data Processing: For each condition and task, the software segmented the foot into anatomical regions (heel, midfoot, forefoot, toes). The values for the entire foot's contact area, average pressure, and peak pressure were exported for statistical analysis.

   3.4. Statistical Analysis The collected data was analyzed using repeated-measures Analysis of Variance (ANOVA) to determine if the differences observed between the four carrying conditions were statistically significant (p < 0.05). Post-hoc tests (Bonferroni correction) were then applied to identify exactly which pairs of conditions were different from each other (e.g., Is unilateral right significantly different from no backpack?).
4. Detailed Results and Biomechanical Interpretation Surface Contact Area: The analysis revealed a significant increase (p<0.05) in the contact area for both feet, but in a specific pattern.

   The right foot contact area increased significantly during bilateral carrying and unilateral right carrying compared to the no-backpack condition.

   The left foot contact area increased significantly during unilateral left carrying.

   Interpretation: The body's primary adaptation to asymmetrical loading is to increase stability by "splaying" the foot, creating a larger base of support. This is a compensatory mechanism to prevent loss of balance. The fact that bilateral carrying also increased contact area on the right foot may suggest a natural limb dominance or subtle postural shifts even under symmetrical load.

   Average and Peak Pressure: Contrary to what might be expected, there were no statistically significant changes in either the average pressure across the foot or the peak (maximum) pressure points under any of the carrying conditions, during both standing and walking.

   Interpretation: This is a critical finding. It demonstrates the remarkable adaptive capacity of the healthy adolescent musculoskeletal system. The body successfully manages the added 15% load not by increasing pressure intensity, but by efficiently redistributing it over a larger surface area. This prevents potentially harmful focal points of high pressure that could lead to pain or tissue damage in the short term. This efficient redistribution is likely achieved through subtle adjustments in muscle activation around the foot, ankle, and leg.

   Bilateral Comparison: During dynamic walking, no significant pressure imbalance was created between the left and right foot across conditions.

   Interpretation: The gait cycle itself acts as a natural equalizer. The rhythmic, alternating pattern of walking appears to mitigate the asymmetrical load imposed during unilateral carrying, preventing a sustained left-right discrepancy in pressure output.
5. Discussion, Limitations, and Future Research Discussion: This study provides quantitative evidence that the body's immediate response to backpack load is a strategic increase in foot contact area to maintain stability, rather than an increase in plantar pressure intensity. While this adaptation is effective, it represents an altered and potentially less efficient biomechanical state. Chronic adoption of a unilateral carrying posture could lead to muscular fatigue, joint stress, and long-term postural alignment issues upstream in the kinetic chain (ankles, knees, hips).

   Limitations:

   The study assessed immediate effects. Long-term longitudinal research is needed to see if these adaptations lead to permanent changes or pathology.

   The participants were healthy. Results may differ in adolescents with pre-existing musculoskeletal conditions.

   The study was conducted barefoot. Footwear would interact with load carriage and is an important area for future study.

   Future Research Directions:

   Investigation of heavier loads (e.g., 20% of body weight) to find a potential "breaking point" of this adaptive mechanism.

   Electromyography (EMG) studies are used to measure which muscles are activated to facilitate this pressure redistribution.

   Long-term studies following adolescents through their school years to correlate carrying habits with the development of pain or postural issues.
6. Conclusion and Practical Recommendations In conclusion, this detailed biomechanical analysis confirms that the backpack carrying method significantly influences adolescent posture at the foundational level. The body compensates for uneven loads intelligently, but this compensation comes at the cost of altered natural foot mechanics.

Evidence-Based Recommendations:

Promote Bilateral Carriage: The consistent use of both shoulder straps is the single most effective way to minimize asymmetric biomechanical adaptations.

Monitor Weight: Strictly adhere to the 10-15% of body weight guideline to remain within the body's effective compensatory range.

Ensure Proper Fit: Backpacks should be positioned high on the back, snug against the body, with the bottom above the waist. The use of hip belts and chest straps should be encouraged to distribute the load more effectively to the pelvis.

Educate on Risks: Adolescents and their parents should be made aware that even if no pain is felt, carrying a backpack on one shoulder can disrupt normal body mechanics and may have long-term consequences.

Incorporate into Clinical Practice: Healthcare providers should include backpack habits in their patient history for adolescents presenting with any lower limb or back pain.

ELIGIBILITY:
Inclusion Criteria:

* • Their age will range from 12 to 18 years.

  * Their body mass index (BMI) is within normal range according to BMI for age percentile score (WHO, 2007).
  * All adolescents will be free from postural deviation, the trunk rotation in all students is within a normal degree determined by scoliometer (Bunnel, 1993).

Exclusion Criteria:

* Visual, auditory, or perceptual deficits.
* Deformities at any joint of the lower limbs and spine.
* Surgical intervention in the foot.
* Deep sensory loss.
* Musculoskeletal disorders.

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: This study will be conducted on ninety-two healthy adolescents from both sexes to determine the effect of different backpack carriage styles on plantar pressure distribution in adolescents. They will be recruited from public and private schools in Mansoura city.
Sampling Method: Non-Probability Sample
Enrollment: 92 (Actual)
Dates: Start 2022-01-15 (Actual); Primary Completion 2023-07-25 (Actual); Study Completion 2023-09-10 (Actual)

PRIMARY OUTCOMES:
Change in the Planar pressure distribution across the foot at different backpack carrying conditions. | 2 Hours
  The plantar pressure distribution was recorded using the Foot Scan Plate System under different conditions, (Maximum pressure-contact surface area-average pressure) were recorded.
  The conditions are:
  1. Without Backpack
  2. Carrying a Backpack with a Unilateral strap on the Left shoulder
  3. Carrying a Backpack with a Unilateral strap on the Right shoulder
  4. Carrying a Backpack with Bilateral straps on both shoulders

CONTACTS AND LOCATIONS:
Locations (1):
- Orthomedics, Al Mansurah, Egypt

IPD SHARING:
Plan to Share IPD: Yes
All IPD collected throughout the trial
Supporting Information: Study Protocol, SAP, ICF

REFERENCES:
- [Background] Pau M, Leban B, Corona F, Gioi S, Nussbaum MA. School-based screening of plantar pressures during level walking with a backpack among overweight and obese schoolchildren. Ergonomics. 2016 May;59(5):697-703. doi: 10.1080/00140139.2015.1077275. Epub 2015 Sep 7. PMID 26226045

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-09-15): https://cdn.clinicaltrials.gov/large-docs/49/NCT07161349/Prot_SAP_000.pdf
  • Informed Consent Form (2023-09-15): https://cdn.clinicaltrials.gov/large-docs/49/NCT07161349/ICF_001.pdf